CLINICAL TRIAL: NCT01902732
Title: Bronchoscopic Volume Reduction With Valve Implants After Analysis of Interlobar Fissure Integrity and Measurement of Collateral Ventilation in Patients With Severe, Heterogeneous Emphysema
Brief Title: Endoscopic Lung Volume Reduction After Catheter-based CV Measurement in Patients With Heterogeneous Emphysema and Complete Interlobar Fissures
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Prof. Dr. med. Felix JF Herth, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol G1.0.- 16.02.2012
Record Dates: First submitted 2013-06-13; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Heterogeneous Emphysema

ARMS (1):
- Implantation of valves (IBV) (Other): Following catheter-based measurement of collaertal ventilation, each patient is treated by a complete occlusion of the targeted lobe by intrabronchial valves.
  Interventions: Device: Implantation of valves (IBV)

INTERVENTIONS:
Device: Implantation of valves (IBV) — Implantation of intrabronchial valves in the most emphysematous destroyed and hyperinflated lung lobe improves the elastic recoisl of the samll airways by a reduction in lung volume and thus leading to more ergonomic breathing mechanics and diaphragm function. This positive effect is observed particularly in patients with low interlobar collateral ventilation that can be quantified by CT fissure analysis and/or catheter-based measurement.
  Other Names: Spiration(R) valves

SUMMARY:
This clinical trial evaluates the impact of catheter-based measurement of interloabr collateral ventilation prior to endoscopic lung volume reduction in patients with hetereogeneous emphysema and complete interlobar fissures in high resolution computed tomography.

DETAILED DESCRIPTION:
50 patients (25 per center) with heterogeneous lung emphysema with indication for endoscopic lung volume reduction by valve implantation will be prospectively included in the study. Heterogeneity of emphysema and fissure completeness of the relevant lobe will be proven from high resolution computed tomography (HRCT) prior to enrolment in the study. Fissure integrity will be analyzed by a core radiology. If fissure completeness is proved, patients will be enrolled in the study. All recruited patients will additionally receive a collateral ventilation measurement by using the Chartis® Pulmonary Assement System during a flexible bronchoscopy. Depending on the results of this measurement, patients are divided in two parallel arms: A: complete fissure integrity and low collateral ventilation (CV negative) B: complete fissure integrity and high collateral ventilation (CV positive) Following the CV measurement, each patient will receive valve therapy.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* ability to understand the importance of adherence to study treatment and the study protocol and willing to follow all study requirements
* severe lung emphysema (FEV1<45%, RV>150%, TLC>100%)
* pO2>60 mmHg with 4l O2, pCO2 < 60 mmHg at rest
* heterogeneous lung emphysema diagnosed with HRCT and perfusion scintigraphy
* confirmed heterogeneity by YACTA®
* disclosure of parallel channels through relevant interlobar fissures
* age > 30 years
* stable COPD without exacerbation 8 weeks prior to screening
* dose of cortisone< 20 mg prednisone or equivalent OCS
* non-smoker or ex-smoker who stopped smoking for at least 4 months prior to the screening visit
* current CoHb < 2,5%

Exclusion Criteria:

* BMI < 18 mg/kg2
* significant bronchiectasis with sputum production of 4 tablespoons/day
* 6-minute-walk distance < 150 m
* myocardial infarction within 6 weeks prior screening visit
* decompensated heart failure
* cardiomyopathy with moderate or severe restricted LVF
* long-term medication with Clopidogrel
* status after lung resection (Lobectomy/Pneumonectomy)
* existing pregnancy
* female subjects of child-bearing potential without acceptable forms of contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Improvement on pulmonary function | 12 months
  Development of lung function parameters FEV1 and RV/TLC. Increase of FEV1 of 15% and decrease of RV/TLC of 10% compared to baseline will be considered as clinically significant.

SECONDARY OUTCOMES:
Assessment of safety and efficacy | 12 months
  Safety:
  * Evaluation of number of serious adverse events related to the treatment
  * Evaluation of migration rate of valve implants
  * Evaluation of technical difficulties during implantation of valves
  Efficacy:
  * average change in lung function (FEV1, IVC, RV, TLC, RV/TLC) 30 , 90, 180 and 365 days after ELVR
  * average change in life quality (SGRQ) and in dyspnoea score (mMRC)
  * average changes in distance of six minute walk test 30, 90, 180 and 365 days after ELVR
  * average changes in physical activity at home, measured with Sensewear®-wristband for three days 30, 90, 180 and 360 days after ELVR
  * echocardiographic/laboratory chemical changes of cardiac function 30, 90, 180 and 365 days after ELVR.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - LungenClinic Grosshansdorf, Großhansdorf
  - Thoraxklinik Heidelberg, Heidelberg
  - Thoraxklinik, Heidelberg